CLINICAL TRIAL: NCT02857998
Title: A Phase I, Open-label, Dose-escalation Study of the Safety and Pharmacokinetics of HMPL-523 in Patients With Relapsed or Refractory Mature B-cell Neoplasms
Brief Title: A Study of Hutchison MediPharma Limited(HMPL)-523 in Patients With Relapsed or Refractory Mature B-cell Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-523-00CH1
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Mature B-cell Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HMPL-523 (Experimental): Oral administration, at dose of 200, 400, 600 and 800 mg once daily;at dose of 200,300, 400mg twice daily at Dose-escalation stage; At Dose-expansion stage, if patients dosing at 600mgQD.
  Interventions: Drug: HMPL-523

INTERVENTIONS:
Drug: HMPL-523 — Oral administration, once daily
  Other Names: HMPL-523 Acetate

SUMMARY:
A Phase I, Open-label, Dose-escalation Study of the Safety and Pharmacokinetics of HMPL-523 in Patients With Relapsed or Refractory Mature B-cell Neoplasms

DETAILED DESCRIPTION:
There are two stages in this study: a dose-escalation stage (stage 1) and a dose-expansion stage (stage 2).

Dose-escalation stage (stage 1):

The conventional 3+3 design (3 patients per dose cohort, with the potential to add additional 3 patients to the same cohort to further evaluate toxicity) will be applied for dose escalation and maximum tolerated dosage determination. Approximately 27 to 42 dose limited toxicities evaluable patients will be enrolled. The actual number of patients depends on the dose limited toxicities situation as well as the maximum tolerated dosage reached at this stage.

Dosing will begin at 200mg once daily. A cycle of study treatment will be defined as 28 days of continuous dosing.

Dose-expansion stage (stage 2):

This phase is to further evaluate the safety, the pharmacokinetics and anti-tumor activity of HMPL-523 at recommended phase 2 dosage in approximately 190 patients with relapsed or refractory Hematologic Malignancies.

In this stage, approximately 190 patients with Mature B-cell Neoplasms will be enrolled with recommended phase 2 dosage 600milligram(mg) one a day(QD) as starting dosing. The tumor types of the expansion stage are restricted to Chronic lymphocytic leukemia/ small lymphocytic lymphoma (CLL/SLL), Mantle cell lymphoma (MCL), Follicular Lymphoma (FL), Diffuse large B-cell lymphoma (DLBCL), Marginal zone lymphoma (MZL)and Waldenstrom's macroglobulinemia (WM)/Lymphoplasmacytic lymphoma(LPL) Subjects will receive HMPL-523 with every 28-day treatment cycle until disease progression, death, or intolerable toxicity, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age >=18 years
3. Histologically relapsed or refractory mature B-cell Neoplasms, have failed at least one prior therapy or patients who are unable to tolerate standard therapy or no curative therapy or therapy of higher priority exists
4. Eastern Cooperative Oncology Group（ECOG） performance status of 0 or 1
5. Expected survival of more than 24 weeks as determined by the investigator
6. In expansion stage, Subjects should have at least one dual diameter measurable lesion expect for subject with CLL or subject with LPL/WM with abonormal immunoglobulin

Exclusion Criteria:

1. Patients with primary central nervous system(CNS) lymphoma
2. Any of the following laboratory abnormalities:

   * Absolute neutrophil count<1.5×109/L
   * Hemoglobin <80g/L
   * Platelet<75 ×109 /L
3. Inadequate organ function, defined by the following:

   * Total bilirubin >1.5the ULN with the following exception:

     * Patients with known Gilbert disease who have serum bilirubin level ≤3 the upper limit of normal(ULN) and normal Aspartate aminotransferase(AST)/Alanine aminotransferase(ALT) may be enrolled.
4. AST and/or ALT > 2.5 the ULN with the following exception:Patients with documented disease infiltration of the liver may have AST and/or ALT levels ≤ 5 the ULN.
5. Serum amylase or lipase > the ULN
6. Serum creatinine > 1.5 the ULN or estimated creatinine clearance < 50 mL/min
7. International normalized ratio (INR)>1.5 the ULN or activated partial thromboplastin time (aPTT)>1.5 the ULN
8. Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, or current known active infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV)
9. Pregnant (positive pregnancy test) or lactating women
10. New York Heart Association (NYHA) Class II or greater congestive heart failure
11. Congenital long QT syndrome or corrected QT interval (QTc) > 480 msec
12. Currently use medication known to cause QT prolongation.
13. Subjects with presence of clinically detectable second primary malignant tumors at enrollment, or other malignant tumors within the last 2 years (with the exception of radically treated basal cell or squamous cell carcinoma of the skin, in situ cervix, or in situ breast cancer).
14. Any anti-cancer therapy, including chemotherapy, hormonal therapy, biologic therapy, or radiotherapy within 3 weeks prior to initiation of study treatment
15. Herbal therapy ≤1 week prior to initiation of study treatment
16. Prior treatment with any spleen tyrosine kinase (SYK) inhibitors (Fostamatinib)
17. Prior allogeneic stem cell transplant within 6 months prior to initiation of study treatment or with any evidence of active graft versus host disease or requirement for immunosuppressants within 28 days prior to initiation of study treatment
18. Clinically significant active infection (pneumonia)
19. Major surgical procedure within 4 weeks prior to initiation of study treatment
20. History of myocardial infarction or unstable angina within 6 months prior to initiation of study treatment
21. Inability to take oral medication, prior surgical procedures affecting absorption, or active peptic ulcer disease
22. Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤1, except for alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Dose limited toxicities evaluated with NCI CTCAE v4.03 | within 28 days after the first dose
  Incidence of dose limited toxicities and associated dose of HMPL-523

SECONDARY OUTCOMES:
Maximum plasma concentration calculated with Blood samples | within 29 days after the first dose
  Blood samples will be taken to measure the levels of study drug
Time to reach maximum concentration calculated with Blood samples | within 29 days after the first dose
  Blood samples will be taken to measure the levels of study drug
Objective response rate | within 30 days after the last dose
  the proportion of subjects who have a Complete Response or Partial Response
Adverse events evaluated by NCI CTCAE v4.03 | from the first dose to within 30 days after the last dose
  Incidence of adverse events and associated dose of HMPL-523

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yang, M.D., Study Chair — Hutchison Medipharma Ltd.
Locations (2):
- China (2):
  - BeijingCancer Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song Y, Cao J, Zhang Q, Li C, Qiu L, Qi J, Zhang H, Li W, Liu L, Jing H, Zhou K, Zhang W, Zhang L, Li D, Zou L, Yang H, Qian W, Zhou H, Hu J, Yin H, Fu S, Fan S, Xu Q, Wang J, Jia X, Dai G, Su W, Zhu J. Phase I study of the Syk inhibitor sovleplenib in relapsed or refractory mature B-cell tumors. Haematologica. 2024 Jul 1;109(7):2165-2176. doi: 10.3324/haematol.2022.282401. PMID 38235512